CLINICAL TRIAL: NCT01387594
Title: A Multi-Center, Phase 1, Open-Label Evaluation Of The Effect Of PF-00547659 (Anti Madcam Monoclonal Antibody) On Cerebrospinal Fluid (CSF) Lymphocytes In Volunteers With Crohns Disease Or Ulcerative Colitis Who Are Anti-TNFInadequate Responders (TOSCA)
Brief Title: Evaluate PF-00547659 On Cerebrospinal Fluid Lymphocytes In Volunteers With Crohn's Disease Or Ulcerative Colitis Who Failed Or Did Not Tolerate Anti-TNFs
Acronym: TOSCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A7281008; 2011-001443-74 (EudraCT Number)
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease; Ileitis; Ileo-colonic and Colonic Crohn's Disease; Granulomatous Colitis; Regional Enteritis; Ulcerative Colitis
Keywords: Crohn's disease lumbar puncture anti-MAdCAM monoclonal antibody PF-00547659 Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Ileitis; Colitis, Ulcerative | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Interventions prior to treatment. Control arm
  Interventions: Procedure: lumbar puncture
- Cohort 2 (Experimental): Interventions prior to and after 3 monthly injections
  Interventions: Drug: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture — 2 lumbar punctures prior to treatment; study drug 225mg SC once a month X 3 doses.
  Arms: Cohort 1
Drug: lumbar puncture — 1 lumbar puncture before and after 3 doses; study drug 225mg SC once a month X 3 doses.
  Arms: Cohort 2

SUMMARY:
Study is designed to show a lack of effect on white blood cells circulating in the spinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* males and females >=18 and =<75 years
* For CD subjects: hsCRP > 5 mg/L and Harvey-Bradshaw Index > 8 OR when HBI cannot be determined (ie if stoma is present) or hsCRP < 5mg/L then: active lesions on colonoscopy or flexible sigmoidoscopy or active Crohn's disease on CT or MR enterography
* For UC subjects: diagnosis of UC > 3 months; must have endoscopy to confirm active disease during screening; total mayo score of 6 to 12 points and moderate to severe disease on endoscopy

Exclusion Criteria:

* Pregnancy or breastfeeding
* TB or active enteric infections
* Entero vesicular fistulae
* Prior use of natalizumab or vedolizumab
* Right or left heart failure including symptomatic diastolic dysfunction or unexplained elevation of troponin I (>0.05 ng/mL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2015-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- AKH Wien Universitaetsklinik fuer Innere Medizin III Klinische Abteilung fuer Gastroenterologie und, Vienna, Austria
- Belgium (2):
  - Hopital Erasme, Brussels
  - UZ Gasthuisberg, Leuven
- France (4):
  - Hopital Cardiologique, Lille
  - Hopital Huriez, CHRU de Lille, Lille
  - Hopital Saint-Louis - CIC, Paris
  - Hopital Saint-Louis, Paris
- Charité, Universitaetsmedizin Berlin, Campus Virchow Klinikum,, Berlin, Germany
- Academic Medical Center - University of Amsterdam, Dept. of Gastroenterology, Amsterdam, Netherlands

REFERENCES:
- [Derived] Stuve O, Cataldi F, Pradhan V, Gorelick KJ. Normal intrathecal leukocyte cell number and composition do not decrease the incidence of post-lumbar puncture headache. J Neuroimmunol. 2017 Sep 15;310:69-71. doi: 10.1016/j.jneuroim.2017.06.011. Epub 2017 Jun 30. PMID 28778448
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281008&StudyName=A%20Multi-center%2C%20Phase%201%2C%20Open-label%20Evaluation%20Of%20The%20Effect%20Of%20Pf-00547659%20%28anti%20Madcam%20Monoclonal%20Antibody%29%20On%20Cerebrospinal%20Fluid%20%28csf%29%20Lymphocytes%20In%20Volunteers%20With%20Crohns%20Disease%20Or%20Ulcerative%20Colitis%20Who%20Are%20Anti-tnf%20Inadequate%20Responders%20%28tosca%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: PF-00547659: Participants who had Crohn's disease (CD) and who satisfied all study entry criteria were enrolled into the study. Prior to treatment, participants underwent 2 lumbar punctures (LP) 2-4 weeks apart. All participants received 3 monthly subcutaneous (SC) doses of PF-00547659 225 milligrams (mg) (Days 1, 29, 57). At Week 12, participants who had a clinical response to treatment could enter the open-label extension study. Otherwise, participants would enter a 6-month follow-up period onsite.
- Cohort 2: PF-00547659: Participants who had Crohn's disease (CD) and who satisfied all study entry criteria were enrolled into the study. Participants underwent 2 lumbar punctures (LP), 1 prior to treatment and another 1-3 weeks after the last dose. All participants received 3 monthly subcutaneous (SC) doses of PF-00547659 225 milligrams (mg) on Days 1, 29, and 57. At Week 12, participants who had a clinical response to treatment could enter the open-label extension study. Otherwise, participants would enter a 6-month follow-up period onsite.
Period: Overall Study
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659
Started | 10 | 39
Completed | 10 | 36
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659 | Total
Number analyzed (Participants) | 10 | 39 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.9) | 37.4 (10.6) | 38.1 (11.8)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 6 | 27 | 33
  45-64 years | 4 | 12 | 16
  More than or equal to (>=) 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 26 | 28
  Male | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cohort 2: Baseline Absolute Lymphocyte Count in Cerebrospinal Fluid (CSF)
Description: The primary CSF endpoint of Cohort 2 was the percent change from baseline in absolute lymphocyte counts in CSF after 3 doses of PF-00547659. The hypothesis for the primary endpoint was evaluated using the CSF evaluable population in Cohort 2. CSF samples were obtained via lumbar puncture and analyzed by fluorescence-activated cell sorting (FACS) for total lymphocyte counts. Lumbar punctures were performed by a highly qualified physician using a 20-22 gauge needle, preferably an atraumatic needle.
Time Frame: Baseline
Population: All Cohort 2 participants who were enrolled, had 2 evaluable LPs, and who received all 3 doses of study drug.
Measure: Median (Full Range); unit: cells per milliliter (cells/mL)
Arm/Group | Cohort 2: PF-00547659
Number analyzed (Participants) | 32
cells per milliliter (cells/mL) | 338.5 (689.69) [67.0 to 2100.0]

2. Primary Outcome: Cohort 2: Percent Change From Baseline in Absolute Lymphocyte Count in CSF at Month 3
Description: The primary CSF endpoint of Cohort 2 was the percent change from baseline in absolute lymphocyte counts in CSF after 3 doses of PF-00547659. The hypothesis for the primary endpoint was evaluated using the CSF evaluable population in Cohort 2. CSF samples were obtained via lumbar puncture and analyzed by FACS for total lymphocyte counts. Lumbar punctures were performed by a highly qualified physician using a 20-22 gauge needle, preferably an atraumatic needle.
Time Frame: Baseline, Month 3
Population: All Cohort 2 participants who were enrolled, had 2 evaluable lumbar punctures, and who received all 3 doses of study drug.
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 2: PF-00547659
Number analyzed (Participants) | 32
percent change | 35.2 (92.67) [-70.2 to 267.8]
Statistical Analysis 1: Comparison: Cohort 2: PF-00547659; The null hypothesis is the (median) percent decrease in total lymphocytes count is greater or equal to 50%, equivalently indicating that the geometric mean ratio (GMR: post-treatment/pretreatment) in total lymphocyte counts is less than or equal to 0.5; Test type: Superiority or Other; A p-value was not computed; hypothesis was tested using confidence interval (CI) approach; Geometric Mean Ratio (GMR) = 1.33, 80% CI 2-sided [1.13 to 1.56] — The lower limit of 80% CI greater than 0.5 indicates the statistical significance at alpha=0.1 level

3. Secondary Outcome: Cohorts 1 and 2: Total Number of Participants With Non-Lumbar Puncture (LP) Related Treatment-Emergent Adverse Events (AEs), Withdrawals Due to AEs, and Serious Adverse Events (SAEs) During the 12-week Treatment Period
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent for this measure are events between first dose of study drug and up to 85 days (Week 12) after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included serious and non-serious AEs.
Time Frame: Baseline up to Week 12
Population: All participants who received at least one dose of study drug were analyzed for AEs/safety. Combined data for both cohorts is presented.
Measure: Number; unit: participants
Groups:
- Cohort 1: PF-00547659: Participants who had CD and who satisfied all study entry criteria were enrolled into the study. All participants received 3 monthly subcutaneous (SC) doses of PF-00547659 225 milligrams (mg) (Days 1, 29, 57). 2 LPs were to be performed during participation. At Week 12, participants who had a clinical response to treatment could enter the open-label extension study. Otherwise, participants would enter a 6-month follow-up period onsite.
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659
Number analyzed (Participants) | 10 | 39
participants
  AEs | 9 | 36
  Withdrawals due to AEs | 0 | 0
  SAEs | 1 | 3

4. Secondary Outcome: Cohorts 1 and 2: Number of Participants Who Developed Anti-Drug Antibodies (ADAs) to PF-00547659
Description: Serum samples were analysed for presence of ADAs to PF-00547659. Participants who showed positive results for PF-00547659 were reported.
Time Frame: Day 1; Weeks 4, 8, 9-11 (Cohort 2 only), 12, 20, 28, and 36; Early Withdrawal
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 1: PF-00547659: Participants who had Crohns disease (CD) and who satisfied all study entry criteria were enrolled into the study. Prior to treatment, participants underwent 2 lumbar punctures (LP) 2-4 weeks apart. All participants received 3 monthly subcutaneous (SC) doses of PF-00547659 225 milligrams (mg) (Days 1, 29, 57). At Week 12, participants who had a clinical response to treatment could enter the open-label extension study. Otherwise, participants would enter a 6-month follow-up period onsite.
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659
Number analyzed (Participants) | 10 | 39
participants | 4 | 11

5. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Injection Site Reactions by Severity
Description: Injection site reaction AEs include: injection site irritation, injection site pain, injection site rash, contusion, and erythema.
Time Frame: Baseline till End of Study/Early Withdrawal, up to Week 12
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659
Number analyzed (Participants) | 10 | 39
participants
  Mild | 1 | 6
  Moderate | 0 | 1
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening till end of study or at early withdrawal, whichever was earlier, up to Week 12.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Cohort 1: PF-00547659 | Cohort 2: PF-00547659
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/39
Other Adverse Events (participants affected / at risk) | 9/10 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-00547659 (N=10) | Cohort 2: PF-00547659 (N=39)
Crohn's disease (Gastrointestinal disorders) | 0 | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-00547659 (N=10) | Cohort 2: PF-00547659 (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Eye inflammation (Eye disorders) | 0 | 2
Eye pain (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 5
Injection site irritation (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 2
Injection site rash (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Celluliitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Herpes ophthalmic (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 1
Laryngitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 7
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Stoma site abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 7
Restless legs syndrome (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Perineal erythema (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Nail pitting (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.